CLINICAL TRIAL: NCT01350297
Title: Phrenic Reinnervation in Central Ventilatory Paralysis Due to Medullary Trauma With Phrenic Motoneuron Destruction
Brief Title: Diaphragmatic Reinnervation of Tetraplegic Patients With Respiratory Insufficiency
Acronym: TETRADIA-UNI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/023/HP
Record Dates: First submitted 2010-02-02; First posted 2011-05-09 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Tetraplegia
Keywords: tetraplegia; reinnervation; phrenic nerve
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Experimental): Patients
  Interventions: Procedure: reinnervation

INTERVENTIONS:
Procedure: reinnervation — anastomosis between right inferior laryngeal nerve and right phrenic nerve
  Other Names: laryngeal reinnervation

SUMMARY:
This study evaluates the diaphragmatic reinnervation by inferior laryngeal nerve in tetraplegic patients with ventilatory insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* tetraplegia c3-c4
* respiratory insufficiency

Exclusion Criteria:

* PM

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
recovery of spontaneous ventilation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: VERIN Eric, MD, Study Chair — University Hospital, Rouen
Locations (1):
- VERIN, Rouen, France